CLINICAL TRIAL: NCT02323789
Title: A Phase I/II Study Evaluating Allogeneic Mesenchymal Stromal Cells in Adults With Recessive Dystrophic Epidermolysis Bullosa
Brief Title: Mesenchymal Stromal Cells in Adults With Recessive Dystrophic Epidermolysis Bullosa
Acronym: ADSTEM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADSTEM001
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Recessive Dystrophic Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention arm (Experimental): 10 patients with RDEB will be selected to receive the intervention - mesenchymal stromal cells.
  Interventions: Drug: Mesenchymal stromal cells

INTERVENTIONS:
Drug: Mesenchymal stromal cells — TC-MSC: a cell product containing mesenchymal stromal cells. Mesenchymal stromal cells are adherent non-haematopoietic multipotent cells that are expanded from bone marrow from healthy donors, using platelet lysate as source of growth factor.
  Other Names: TC-MSC

SUMMARY:
To assess whether intravenously administered third-party bone marrow-derived mesenchymal stromal cells (MSCs) are safe and have an impact on disease severity in RDEB

DETAILED DESCRIPTION:
This is a phase I/II clinical trial with a key objective of evaluating safety of third party bone MSCs intravenous infusions in 10 adults with the inherited severe skin fragility disorder, recessive dystrophic epidermolysis bullosa (RDEB). The main objectives of our study are to: (1) to assess the spectrum of clinical responses in adults with RDEB receiving intravenous MSCs; (2) to identify the best cohort of individuals to target for future trials and therapies; (3) to improve our understanding of in vivo and in vitro responsiveness to MSCs; (4) to identify candidate molecules germane to activating MSCs and making them clinically more potent, independently of the permissive conditions of the patient and (5) to assess its impact on reducing disease morbidity/severity in this population.

This is a prospective, non-randomised, open label study. All study participants will receive two intravenous MSC infusions at baseline Day 0 and Day 14 and will be followed up for a 12 month period following the first infusion. Each subject will undergo an initial screening including physical examination, assessment of vital signs and disease severity assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with a diagnosis of RDEB confirmed by DNA analysis and skin immunofluorescence for partial or complete absence of type VII collagen.
2. Individuals ≥ 18 years and ≤ 65 years of age, both male and female
3. Individuals that have voluntarily signed and dated an informed consent form (ICF) prior to the first study intervention.

Exclusion Criteria:

1. Subjects who have had other investigational medicinal products within 90 days prior to screening or during the treatment phase.
2. Subjects who have received immunotherapy including oral corticosteroids for more than 1 week (intranasal and topical preparations are permitted).
3. Subjects with a known allergy to any of the constituents of the investigational product.
4. Subjects with a medical history or evidence of malignancy, including cutaneous squamous cell carcinoma.
5. Subjects who are pregnant or of child-bearing potential who are not abstinent or practicing an acceptable means of contraception, as determined by the Investigator, for the duration of the treatment phase.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Lack of serious and severe adverse events (SAEs) related to the administration of the investigational medicinal product. | 12 months

SECONDARY OUTCOMES:
Presence of new type VII collagen at the dermal-epidermal junction post treatment. | Day 14, Day 28, Day 60, Day 100 and Month 6.
Change in general markers of inflammation | Day 14, Day 28, Day 60, Day 100, Month 6 and Month 12 compared to baseline
Changes in specific markers of inflammation | Day 14, Day 28, Day 60 and Month 6 compared to baseline
Change in the clinical changes in the skin assessed with clinical photographs | Day 14, Day 28, Day 60, Day 100, Month 6 and Month 12.
Differences in quality of life data | Day 28, Day 60, Day 100, Month 6 and Month 12 compared to baseline
Change in BEBSS and EBDASI scores | at Day 28, Day 60, Day 100, Month 6 and Month 12 compared to baseline
Change in Pain scores | Day 28, Day 60, Day 100, Month 6 and Month 12 compared to baseline
Change in pruritus score using the Leuven Itch Scale (LIS) | Day 28, Day 60, Day 100, Month 6 and Month 12 compared to baseline.
Quantification of total blister numbers over the entire body surface area | Day 28, Day 60, Day 100, Month 6 and Month 12 compared to baseline
10. Increase in the skin strength measured by time to blister formation after negative pressure skin suction test | Day 28, Day 60, Day 100, Month 6 and Month 12 compared to baseline
Qualitative analyses based on a series of interview questions | between screening and Day 0, between Day 28 and Day 60, and between Month 6 and Month 12.
  to reveal objective data on quality of sleep, skin healing time, amount of dressings used, improvement in oral diet, improvement in energy levels, mood, quality of family life/relationships.

CONTACTS AND LOCATIONS:
Overall Officials: John McGrath, FRCP/FSci/MD, Principal Investigator — King's College London
Locations (1):
- Guys and St Thomas' hospital NHS Trust, London, United Kingdom